CLINICAL TRIAL: NCT03568812
Title: The Role of Probiotics L. Plantarum, S. Thermophiles, B. Bifidum on Gut Inflammation, Bacterial Translocation, and CD4+ Cell Count in HIV Patients With Immunological Non-Responder
Brief Title: The Role of Probiotics in HIV Patients With Immunological Non-Responder
Acronym: PIONIR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Erni J. Nelwan, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-10-1001
Record Dates: First submitted 2018-05-14; First posted 2018-06-26 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections; Immunological Abnormality
Keywords: HIV; immunological non responder; gut inflammation
MeSH Terms: conditions — HIV Infections | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: double blind placebo control study
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics Rillus® (Experimental): Rillus®, Chewing tablet containing viable cell 1.0 x 10^9 colony forming unit (Lactobacillus plantarum 8.55 mg, Streptococcus thermophilus 8.55 mg, Bifidobacterium bifidum 2.55 mg, fructooligosaccharide 480 mg), isomalt, xylitol, milk flavour, vanilla flavour Dosage: 1 chewing tablet Frequency: once daily every night Duration: 12 weeks
  Interventions: Drug: Rillus®
- Placebo (Placebo Comparator): Placebo: Chewing tablet with identical flavour, colour, smell, and size as investigational drug Dosage: 1 chewing tablet Frequency: once daily every night Duration: 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rillus® — Eligible subjects will be divided into 2 groups randomly (Rillus® or placebo). The colour, smell, flavour, and size of the chewing tablet are the same between active and placebo drugs. Subjects will consume the tablet once daily at night for 12 weeks.
  Other Names: Rillus® Treatment group
  Arms: Probiotics Rillus®
Other: Placebo — Eligible subjects will be divided into 2 groups randomly (Rillus® or placebo). The colour, smell, flavour, and size of the chewing tablet are the same between active and placebo drugs. Subjects will consume the tablet once daily at night for 12 weeks.
  Other Names: Control group
  Arms: Placebo

SUMMARY:
This study will address HIV patients who are on antiretroviral treatment (ART) and experiencing immunological failure. The cause of immunological failure in HIV patients could be due to several factors such as age, gender, Cluster of Differentiation (CD4)+ count before started treatment and some inflammation in the gut. The C-C Chemokine Receptor 5 (CCR5) receptor on T lymphocyte CD4+ are abundantly found in the gut and attacked by HIV virus during acute infection causing irreversible damage.

The disruption of gut integrity and chronic inflammation further causing translocation of bacteria in gut lumen to the blood. Thus resulting persistent low CD4+ or immunological failure.

This evaluation plan is designed to establish the role of investigation product (probiotics) to improve gut inflammation in HIV patients.

DETAILED DESCRIPTION:
HIV patients could develop immunological failure despite being treated with antiretroviral therapy (ART). Thus resulting the increase of morbidity and mortality among HIV patients, especially in Indonesia. The immunological failure is associated with decreased gut integrity and immunity, increased gut inflammation, and gut bacterial translocation to the blood. Memory CD4+ T cell damage in gut associated lymphoid tissue (GALT) by HIV-1 virus leads to decreased production of Th17 in gut mucosal layer. Furthermore, low level of Th17 facilitates bacterial translocation in HIV patients.

Probiotic supplementation (Lactobacillus) could decrease the gut inflammation in some diseases including HIV infection; thus helps increasing the gut integrity and immunity by repairing the gut mucosal tight junction, increasing mucin production, and regulating gut Th17. As a result, the gut inflammation and bacterial translocation decreases. Nevertheless, the benefit in HIV patients with immunological non responder status has not been established.

The investigators plan to perform double blind randomized clinical trial of probiotics (containing Lactobacillus plantarum, Streptococcus thermophiles, Bifidobacterium bifidum) in HIV patients with immunological non responder status. The Subject who fulfill inclusion criteria, willing to participate and sign informed consent will be randomized into two groups: the group receiving probiotics (n=40) and the group of placebo (n=40). Intervention will be held for 12 weeks. This study will evaluate the gut mucosal integrity and immunity by Th17 measurement; bacterial translocation by 16S ribosomal RNA (16S RNA) measurement; and gut inflammation by fecal calprotectin measurement before and after the intervention. Moreover, the investigators will measure the CD4+ level to assess immune status recovery before and after the intervention. Side effects, HIV symptom index, Food Frequency Questionnaire will also be assessed every 4 weeks.

Statistical analysis will uses: paired and independent t test (if normally distributed) or using Wilcoxon and Mann Whitney test (if not normally distributed). HIV symptom index and Food frequency will be reported descriptively.

ELIGIBILITY:
Inclusion Criteria:

* HIV patient with immunological non-responder status which defined as:
* first line antiretroviral therapy (ART) treated for minimal 6 months
* CD4+ level between 200-410 cell/μL
* HIV viral load <34 copies/mL
* giving consent to participate the study

Exclusion Criteria:

* being pregnant
* lactating
* known Lactobacillus allergy
* BMI <16 kg/m2
* under Tuberculosis treatment or other acute illness
* acute diarrhea
* routinely taking selenium containing vitamin in last 1 month
* routinely consuming probiotics containing product in last 1 month

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erni J Nelwan, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- HIV Clinic, Cipto Mangunkusumo Hospital, Jakarta, Indonesia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was done between May and August 2018, study observation was done for 90-day for each subject and completed in October 2018. During study period patient was recruited consecutively on the day of policlinic visit by evaluate the existing medical record data included (1) data of CD4+ T cell and (2) viral load data at least one year ago (3) using ARV for at least 6-month.
Pre-assignment Details: Eligible patient was offered and signed informed consent while agree to participate. Total of 1771 patients visited POKDISUS. Completed data was available for 111 patients and 80 patients gave informed consent to participate.
Period: Overall Study
Arm/Group | Probiotics Rillus® | Placebo
Started | 40 | 40
Completed | 40 | 39
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotics Rillus® | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (6.7) | 38.2 (6.5) | 39.5 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 29 | 28 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Ambon | 2 | 0 | 2
  Race/Ethnicity: Batak | 2 | 2 | 4
  Race/Ethnicity: Betawi | 4 | 6 | 10
  Race/Ethnicity: Javanese | 16 | 14 | 30
  Race/Ethnicity: Makassar | 1 | 1 | 2
  Race/Ethnicity: Padang | 0 | 3 | 3
  Race/Ethnicity: Palembang | 1 | 0 | 1
  Race/Ethnicity: Riau | 0 | 1 | 1
  Race/Ethnicity: Sumatran | 2 | 0 | 2
  Race/Ethnicity: Sundanese | 3 | 5 | 8
  Race/Ethnicity: Chinese | 7 | 4 | 11
  Race/Ethnicity: Other | 2 | 4 | 6
Th17 Level [Median (Inter-Quartile Range); unit: cell/μL] | 1.4 [0.7 to 2.8] | 1.6 [1.1 to 2.4] | 1.5 [0.8 to 2.4]
CD4+ level [Median (Inter-Quartile Range); unit: cell/μL] | 265 [197 to 394] | 389 [255 to 496.8] | 327 [232 to 436.3]
Fecal Calprotectin Level [Median (Inter-Quartile Range); unit: μg/g] | 6.4 [2.9 to 21.1] | 6.1 [2.6 to 16.1] | 6.3 [2.9 to 16.5]

OUTCOME MEASURES:

1. Primary Outcome: CD4+ Level
Description: CD4 level in blood (cell/μL) indicate immune status of patient receiving probiotics or placebo, measure between baseline and at 12 weeks of intervention. Analysis will include CD4 T cell levels after intervention, adjusted with duration of ARV therapy and baseline CD4 levels, as well as unadjusted.
Time Frame: 12 weeks
Population: The results was divided in to unadjusted and adjusted CD4 level change
Measure: Median (95% Confidence Interval); unit: cell/μL
Arm/Group | Probiotics Rillus® | Placebo
Number analyzed (Participants) | 40 | 39
cell/μL
  The result of unadjusted CD4 level change | 162.3 [112.5 to 212.1] | 50.5 [0.5 to 100.9]
  The result of adjusted CD4 level change | 143.3 [96.9 to 189.7] | 69.9 [22.9 to 117.0]
Statistical Analysis 1: Comparison: Probiotics Rillus® vs Placebo; The statistical analysis of unadjusted CD4 level; Test type: Superiority; p = 0.02, ANCOVA — The threshold for statistical significance was p = 0.05 The variable was adjusted to duration of ARV regimen and baseline CD4 level; Mean Difference (Net) = 111.8, 95% CI 2-sided [40.9 to 182.7] — Treatment difference = Probiotics - Placebo
Statistical Analysis 2: Comparison: Probiotics Rillus® vs Placebo; The statistical analysis of adjusted CD4 level; Test type: Superiority; p = 0.03, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 73.4, 95% CI 2-sided [5.9 to 140.8] — Treatment difference = Probiotics - Placebo

2. Secondary Outcome: Th17 Level Change
Description: Change in Th17 level in blood to assess improvement of gut mucosal integrity and immunity between baseline and at 12 weeks, measured in cell/μL The results was divided in to unadjusted and adjusted Th17 level change.
Time Frame: 12 weeks
Population: The results was divided in to unadjusted and adjusted Th17 level change
Measure: Median (95% Confidence Interval); unit: cell/μL
Arm/Group | Probiotics Rillus® | Placebo
Number analyzed (Participants) | 40 | 39
cell/μL
  The results of unadjusted Th17 level change | -0.5 [-1.0 to 0.1] | -0.2 [-1.8 to 0.3]
  The results of adjusted Th17 level change | -0.3 [-0.8 to 0.2] | -0.4 [-0.9 to 0.1]
Statistical Analysis 1: Comparison: Probiotics Rillus® vs Placebo; The statistical analysis of unadjusted Th17 change after intervention; Test type: Superiority; p = 0.55, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.5 to 1.0] — There is no difference between probiotics - placebo
Statistical Analysis 2: Comparison: Probiotics Rillus® vs Placebo; The statistical analysis of adjusted Th17 change after intervention; Test type: Superiority; p = 0.79, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.7 to 0.9] — There is no difference between probiotics - placebo

3. Secondary Outcome: 16S Ribosomal RNA (rRNA) Total
Description: Total of 16SrRNA of translocated gut bacteria in blood, measured in copies/mL, presented as median and interquartile range.
Time Frame: 12 weeks
Population: 16S rRNA gene level was measured in all participant before and after intervention. The results were undetected in all participants.
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Probiotics Rillus® | Placebo
Number analyzed (Participants) | 40 | 39
copies/mL | NA [NA to NA] — All results are under detection limit. | NA [NA to NA] — All results are under detection limit.

4. Secondary Outcome: Fecal Calprotectin Level Change
Description: Change in calprotectin level in feces to assess gut inflammation between baseline and at 12 weeks, measured in μg/g.
  The results was divided in to unadjusted and adjusted fecal calprotectin level change
Time Frame: 12 weeks
Population: The results are divided in to unadjusted and adjusted fecal calprotectin level change
Measure: Median (95% Confidence Interval); unit: μg/g
Arm/Group | Probiotics Rillus® | Placebo
Number analyzed (Participants) | 40 | 39
μg/g
  The result of unadjusted fecal calprotectin level change | -4.3 [-12.3 to 3.6] | 8.4 [0.4 to 16.3]
  The result of adjusted fecal calprotectin level change | -5.8 [-14.0 to 2.4] | 9.9 [1.6 to 18.1]
Statistical Analysis 1: Comparison: Probiotics Rillus® vs Placebo; The statistical analysis of unadjusted Fecal Calprotectin Level change after intervention; Test type: Superiority; p = 0.03, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -12.7, 95% CI 2-sided [-23.9 to -1.5] — Treatment difference = Probiotics - Placebo
Statistical Analysis 2: Comparison: Probiotics Rillus® vs Placebo; The statistical analysis of adjusted Fecal Calprotectin Level change after intervention; Test type: Superiority; p = 0.01, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -15.6, 95% CI 2-sided [-27.6 to -3.6] — Treatment difference = Probiotics - Placebo

5. Secondary Outcome: Amount of Participants With HIV Related Symptoms
Description: A questionnaire called HIV Symptoms Index (Have been validated in Indonesian language) containing self administered 20 questions consisted of 15 somatic and 5 psychological symptoms to assess Human Immunodeficiency Virus (HIV) related symptoms in patients. The total score is calculated by summing the numbers of each symptom (0 = no symptoms, 1 = no disturbing symptoms, 2 = there are symptoms that are a little annoying, 3 = there are disturbing symptoms, 4 = there are very disturbing symptoms), with a minimum score of 0 and maximum 80. Somatic symptoms range from 0-60 and psychological symptoms range from 0-20. An increase in score indicates a worsening condition. Change in HIV Symptoms Index score to assess improvement of somatic and psychological symptoms between baseline and at 12 weeks.
  The results was divided into somatic and psychological symptoms. Both of them were divided again into unadjusted and adjusted HIV Symptoms Index score Change.
Time Frame: 0,4,8,12 weeks
Population: The results was divided into somatic and psychological symptoms. Both of them were divided again into unadjusted and adjusted HIV Symptoms Index score Change.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Probiotics Rillus® | Placebo
Number analyzed (Participants) | 40 | 39
score on a scale
  The results of unadjusted somatic HIV Symptoms Index score Change | -1.6 [-3.2 to 0.04] | -1.3 [-2.9 to 0.3]
  The results of adjusted somatic HIV Symptoms Index score Change | -1.4 [-2.9 to 0.2] | -1.11 [-2.76 to 0.55]
  The results of unadjusted psychological HIV Symptoms Index score Change | -0.6 [-1.2 to 0.09] | -0.1 [-0.8 to 0.5]
  The results of adjusted psychological HIV Symptoms Index score Change | -0.6 [-1.3 to 0.03] | 0.05 [-0.7 to 0.6]

6. Other Pre Specified Outcome: Change in Food Frequency
Description: Food Frequency Questionnaire (FFQ): A questionnaire consisted of food and drink list and frequency to assess patients' dietary pattern in the past one week. Nutritionist will be asking the participants for the questionnaire questions. The food frequency scaled to "more than one time daily", "once daily", "3-6 times in one week", "1-2 times in one week", "less than one time in one week", "never". We assessed changes in tempeh consumption (as part of FFQ question) after the 12-week intervention by categorizing participants into two groups based on their post-intervention intake: 'seldom' (consuming tempeh 1-2 times per week) and 'often' (consuming tempeh daily). The number of participants in each category was then recorded.
Time Frame: 0,4, 8, 12 weeks
Population: The food frequency is divided in to 2 categories "often and seldom" consume "tempeh" after 12 weeks.
Measure: Number; unit: participants
Arm/Group | Probiotics Rillus® | Placebo
Number analyzed (Participants) | 40 | 39
participants
  consume tempeh 1-2 times in one week. | 22 | 23
  consume tempeh once a day. | 13 | 10
Statistical Analysis 1: Comparison: Probiotics Rillus® vs Placebo; The statistical analysis of food frequency change after intervention (12 weeks); Test type: Superiority; p = 0.551, Chi-squared — The threshold for statistical significance was p = 0.05

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Probiotics Rillus® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotics Rillus® (N=40) | Placebo (N=40)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
This study did not assess the viability of probiotics which were administered through the evaluation of the storage during this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03568812/Prot_SAP_002.pdf
  • Informed Consent Form: Informed Consent Form (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03568812/ICF_001.pdf